CLINICAL TRIAL: NCT04621123
Title: Convalescent Methylene Blue Treated (MBT) Plasma for Early Treatment in Non-hospitalised Mild or Moderate COVID-19 Patients: a Randomized Double Blind Study (COnV-ert)
Brief Title: Plasma for Early Treatment in Non-hospitalised Mild or Moderate COVID-19 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); IrsiCaixa (Other); Banc de Sang i Teixits (Other); Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COnV-ert
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV-2 Infection; Safety and Efficacy
Keywords: Convalescent anti-SARS-CoV-2 MBT Plasma; Convalescent plasma; SARS-CoV-2; Safety; Efficacy
MeSH Terms: conditions — COVID-19 | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective, randomized (1:1), double blind study of Convalescent anti-SARS-CoV-2 MBT Plasma (also known as convalescent plasma) plus standard medical treatment (SMT) versus placebo plus SMT in mild or moderate COVID-19 patients who are non-hospitalised. Subjects will be followed up to 60 days after infusion
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Subjects randomized to convalescent anti-SARS-CoV-2 MBT plasma plus SMT will receive one infusion of 200 to 300 ml of ABO-compatible convalescent plasma obtained from a convalescent donor.
  Interventions: Biological: Convalescent anti-SARS-CoV-2 MBT plasma
- Control Group (Placebo Comparator): Subjects randomized to placebo plus SMT will receive one infusion of 200 to 300 ml of sterile saline solution 0.9%.
  Interventions: Other: Control Group

INTERVENTIONS:
Biological: Convalescent anti-SARS-CoV-2 MBT plasma — Subjects randomized to combination convalescent anti-SARS-CoV-2 MBT plasma plus SMT will undergo an ABO compatibility test and will receive a single infusion of 200 to 300 ml of ABO-compatible convalescent plasma
  Arms: Experimental group
Other: Control Group — Subjects randomized to placebo plus SMT will receive one infusion of 200 to 300ml of sterile saline solution 0.9%.
  Other Names: Sterile saline solution 0.9%
  Arms: Control Group

SUMMARY:
This is a prospective, randomized (1:1), double blind study of Convalescent anti-SARS-CoV-2 MBT Plasma (also known as convalescent plasma) plus standard medical treatment (SMT) versus placebo plus SMT in mild or moderate COVID-19 patients who are non-hospitalised. Subjects with confirmed infection by SARS-CoV-2 will receive SMT plus a total of 200-300 mL of convalescent plasma that has been pathogen-inactivated using MBT or placebo.

Approximately 474 individuals will be randomized (1:1) with an interim analysis after the first 60 subjects (30 in each arm).

The sample size will be re-assessed upon interim analysis. Approximately 135 individuals from selected study sites will be included in the substudy to assess the immune response and the methods of sampling.

This is a prospective, randomized (1:1), double blind study of Convalescent anti-SARS-CoV-2 MBT Plasma (also known as convalescent plasma) plus standard medical treatment (SMT) versus placebo plus SMT in mild or moderate COVID-19 patients who are non-hospitalised. Subjects with confirmed infection by SARS-CoV-2 will receive SMT plus a total of 200-300 mL of convalescent plasma that has been pathogen-inactivated using MBT or placebo.

Approximately 474 individuals will be randomized (1:1) with an interim analysis after the first 60 subjects (30 in each arm).

The sample size will be re-assessed upon interim analysis. Approximately 135 individuals from selected study sites will be included in the substudy to assess the immune response and the methods of sampling.

The investigational product will be administered by IV infusion at baseline. Participants will continue their standard medical treatment (SMT) for SARS-CoV-2 infection as prescribed by their regular physician. If applicable, SMT may be modified during the study, depending on personal requirements, the severity and progression of the disease, and need for hospitalization.

Subjects' participation (from inclusion/baseline visit to the end-of-study visit) will be up to 60 days.

DETAILED DESCRIPTION:
This is a prospective, randomized (1:1), double blind study of Convalescent anti-SARS-CoV-2 MBT Plasma (also known as convalescent plasma) plus standard medical treatment (SMT) versus placebo plus SMT in mild or moderate COVID-19 patients who are non-hospitalised. Subjects with confirmed infection by SARS-CoV-2 will receive SMT plus a total of 200-300 mL of convalescent plasma that has been pathogen-inactivated using MBT or placebo.

Study candidates will voluntarily express their interest in participating in the study through the study website or will be offered to participate at the emergency (ER) and out-patient departments (OPD) of the participating hospitals. Candidates registered on the website will be contacted by study physicians by phone to inform them about the study and check their suitability for the study. Suitable candidates will be scheduled an inclusion/baseline visit in which informed consent will be obtained (i.e., the paper informed consent will be signed), and their eligibility will be confirmed. Candidates identified through ER and OPD departments will undergo an inclusion/baseline visit, where the informed consent will be obtained and eligibility will be checked. A subgroup of eligible candidates from selected study sites will be offered participation in the substudy to assess the immune response and the methods of sampling.

Blood and nasopharyngeal samples will be obtained from all eligible candidates. Eligible candidates will be randomized and administered an intravenous (IV) infusion at baseline (convalescent plasma or placebo). Both the investigator and the participant will be blinded to the study treatment.

Specifically, subjects randomized to combination convalescent anti-SARS-CoV-2 MBT plasma plus SMT will undergo an ABO compatibility test and will receive a single infusion of 200 to 300 ml of ABO-compatible convalescent plasma. Subjects randomized to placebo plus SMT will receive a single infusion of 200 to 300 ml of sterile saline solution 0.9%. Infusion will be administered at baseline, using standard procedures for administration of fresh frozen plasma. Small adults weighing less than 45 kg will receive one infusion of 5 ml of convalescent plasma or placebo per kilogram of body weight.

Participants will be trained on the completion of symptoms diary card and safety diary card.

The participants of the substudy will be drawn an extra tube of blood sample and will be trained on self-collection of middle turbinate (MT) swabs and saliva, and self-collected samples will be obtained.

The symptoms and safety diary card will be filled by the participants daily from baseline to day 14. On follow-up visits on days 3, 7, 14, and 28, all participants will be assessed for clinical and safety outcomes. These visits will be all by telephone except for the day 7 and day 28 visits that will be at home and at hospital, respectively, where additionally blood samples (only on day 7) and nasopharyngeal swabs will be collected.

At day 60 visit, all participants will be assessed by telephone for health-status outcome.

For the participants of the substudy, on day 7, an extra tube of blood sample will be obtained and they will be asked to self-collect MT swabs and saliva. And on day 60, an extra tube of blood sample will be obtained during an additional home or hospital visit.

Approximately 474 individuals will be randomized (1:1) with an interim analysis after the first 60 subjects (30 in each arm).

The sample size will be re-assessed upon interim analysis. Approximately 135 individuals from selected study sites will be included in the substudy to assess the immune response and the methods of sampling.

The investigational product will be administered by IV infusion at baseline. Participants will continue their standard medical treatment (SMT) for SARS-CoV-2 infection as prescribed by their regular physician. If applicable, SMT may be modified during the study, depending on personal requirements, the severity and progression of the disease, and need for hospitalization.

Subjects' participation (from inclusion/baseline visit to the end-of-study visit) will be up to 60 days.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Adult male or female individuals of ≥50 years old.
2. 2. In women of childbearing potential1, negative pregnancy test at inclusion/baseline.
3. 3. Has confirmed SARS-CoV-2 infection as determined by PCR or validated antigen rapid diagnostic test2 from nasopharyngeal swabs ≤5 days prior to inclusion/baseline visit.
4. 4. Symptomatic with mild or moderate COVID-19 with symptoms onset date ≤ 7 days prior to inclusion/baseline visit.

   1. a. Mild COVID-19: Individuals who have any of the common signs and/or symptoms of COVID-19 (i.e., fever, cough, sore throat, malaise, headache, muscle pain) without shortness of breath, dyspnoea, or abnormal chest imaging.
   2. Moderate COVID-19: Individuals who have evidence of lower respiratory disease by clinical assessment or imaging and a saturation of oxygen (SpO2) ≥94% on room air at sea level.
5. 5. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
6. 6. Has understood the information provided and capable of giving informed consent.

1 A woman will be considered of childbearing potential if not permanently sterilized nor postmenopausal. Permanent sterilization methods include tubal ligation, hysterectomy and bilateral oophorectomy. Postmenopausal is defined as 12 months with no menses without an alternative medical cause.

2 PanbioTM COVID-19 Ag Rapid Test (Abbott), STANDARDTM Q COVID-19 Ag Test (Roche) or any other CE marketed test for SARS-CoV-2 Ag detection.

Exclusion Criteria:

1. If female, pregnant, breastfeeding, or planning a pregnancy during the study.
2. Severe or critical COVID-19:

   1. Severe COVID-19: respiratory frequency >30 breaths per minute, SpO2 <94% on room air at sea level, ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mmHg, or lung infiltrates >50%.
   2. Critical COVID-19: respiratory failure, septic shock, and/or multiple organ dysfunction.
3. Current hospital admission for any cause.
4. History of previous confirmed SARS-CoV-2 infection.
5. History of significantly abnormal liver function (Child Pugh C).
6. History of chronic kidney disease (CKD) ≥ stage 4, or need of dialysis treatment.
7. Any pre-existing condition that increases risk of thrombosis.
8. History of allergic reactions to blood or plasma products or methylene blue.
9. Known IgA deficiency with anti-IgA antibodies.
10. Medical conditions for which 300ml of intravenous fluid is considered dangerous (i.e., decompensated heart failure or renal failure with fluid overload).
11. Inability to consent and/or comply with study requirements, in the opinion of the investigator.
12. Currently participating or planning to participate in any interventional study for the treatment of COVID-19 or SARS-CoV-2 infection until day 60.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Hospitalization rate (safety and efficacy) | Day 28
  Assess the therapeutic potential of early administration of convalescent MBT plasma in reducing the rate of hospitalization in non-hospitalised mild or moderate COVID-19 patients.
SARS-CoV-2 viral load (safety and efficacy) | Day 7
  Assess the therapeutic potential of early administration of convalescent MBT plasma in reducing SARS-CoV-2 viral load at day 7, measured by quantitative RT-PCR (RT-qPCR) in non-hospitalised mild or moderate COVID-19 patients.

SECONDARY OUTCOMES:
COVID-19 WHO Clinical progression scale score (safety and efficacy) | Day 60
  Change in COVID-19 World Health Organization WHO Clinical progression scale score to assess hospitalization rate (i.e. who reach a score ≥4).
  * Minimum to maximum scores below:
  * Score 0 (uninfected) - Uninfected; no viral RNA detected
  * Score 1 (ambulatory mild disease) - Asymptomatic; viral RNA detected
  * Score 2 (ambulatory mild disease) - Symptomatic; independent
  * Score 3 (ambulatory mild disease) - Symptomatic; assistance needed
  * Score 4 (hospitalised: moderate disease) - Hospitalised; no oxygen therapy
  * Score 5 (hospitalised: moderate disease) - Hospitalised; oxygen by mask or nasal prongs
  * Score 6 (hospitalised: severe diseases) - Hospitalised; oxygen by NIV or high flow
  * Score 7 (hospitalised: severe diseases) - Intubation Score 8 (hospitalised: severe diseases) - Mechanical ventilation pO2/FiO2 <150 (SpO2/FiO2 <200) or vasopressors
  * and mechanical ventilation, pO2/FiO2 ≥150 or SpO2/FiO2 ≥200
COVID-19 symptoms severity score (safety and efficacy) | Day 14
  Change in COVID-19 symptoms severity score, assessed with the COVID-19 daily self-score tool (FLU- patient-reported outcome measure (FLU-PRO©) PLUS instrument), certified-Spanish translation. COVID-19 daily self-score tool to assess symptom severity across six body systems: nose, throat, eyes, chest/respiratory, gastrointestinal, and body/systemic. Data on the presence/absence of symptoms, symptom profiles, and change over time.
  Items 1-27 are Likert scale questions to score symptom severity (rated 0-4): 0=not at all;4=very much. Items 28-32 are also Likert scale questions (rated 0-4) measuring frequency of specific daily symptoms: 0=never or 0 times;4=always or 4 times. Items 33 and 34 measure the presence/absence of COVID-19 specific symptoms: 0=no;1=yes. Total maximum score of FLU-PRO© PLUS 134
Resolution of symptoms (safety and efficacy) | Day 28
  Time to complete resolution of symptoms
Death rate (safety and efficacy) | Day 60
  Death rate
Adverse events (AE) (safety and efficacy) Adverse events (AE) Adverse events (AE) | Day 28
  Proportion of patients with adverse events (AE) and proportion of grade ≥4 AE, based on the FDA Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers scale
Ferritin (safety and efficacy) | Baseline and Day 7
  Change in inflammatory prognostic markers (ferritin)
Prealbumin (safety and efficacy) | Baseline and Day 7
  Change in inflammatory prognostic markers (prealbumin)
Interleukin 6 (IL-6) (safety and efficacy) | Baseline and Day 7
  Change in inflammatory prognostic markers (Interleukin 6 (IL-6))
D-dimer (safety and efficacy) | Baseline and Day 7
  Change in inflammatory prognostic markers (D-dimer)
C reactive protein (CRP) (safety and efficacy) | Baseline and Day 7
  Change in inflammatory prognostic markers (C reactive protein (CRP))
Leukocyte count (safety and efficacy) | Baseline and Day 7
  Change in inflammatory prognostic markers (Leukocyte count)
Lymphocyte count (safety and efficacy) | Baseline and Day 7
  Change in inflammatory prognostic markers (Lymphocyte count)
Absolute neutralization titers against SARS-CoV-2 in plasma (safety and efficacy) | Baseline and Day 7
  Intergroup comparison of absolute neutralization titers against SARS-CoV-2 in plasma in a subgroup of 135 participants
Titers of neutralizing antibodies against SARS-CoV-2 in plasma (safety and efficacy) | Baseline and Day 60
  Change in titers of neutralizing antibodies against SARS-CoV-2 in plasma in a subgroup of 135 participants
SARS-CoV-2 viral load of self-collected middle turbinate (MT) swab and saliva samples compared to nasopharyngeal swabs collected by a healthcare worker (safety and efficacy) | Baseline and Day 7
  Agreement and SARS-CoV-2 viral load of self-collected middle turbinate (MT) swab and saliva samples compared to nasopharyngeal swabs collected by a healthcare worker in a subgroup of 135 participants
  Outcome 18: Secondary Outcome Measure:
Reduction of SARS-CoV-2 viral load (safety and efficacy) | Baseline and Day 28
  Reduction of SARS-CoV-2 viral load in nasopharyngeal swabs at day 28 after start of treatment, as determined by RT-qPCR

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Hospital Sant Bernabé (Hospital de Berga), Berga, Barcelona
  - CUAP Manresa (Planta 0 del CAP Bages), Manresa, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona

REFERENCES:
- [Derived] Alemany A, Ouchi D, Pradenas E, Aguilar R, Vidal M, Jimenez A, Millat-Martinez P, Corbacho-Monne M, Suner C, Bassat Q, Baro B, Moncunill G, Mitja O; COnV-ert Group of Authors; Blanco J, Dobano C. Patient and donor antibody profiles in early COVID-19 convalescent plasma therapy in the COnV-ert trial. Front Immunol. 2025 Sep 25;16:1647488. doi: 10.3389/fimmu.2025.1647488. eCollection 2025. PMID 41080591
- [Derived] Millat-Martinez P, Gharbharan A, Alemany A, Rokx C, Geurtsvankessel C, Papageorgiou G, van Geloven N, Jordans C, Groeneveld G, Swaneveld F, van der Schoot E, Corbacho-Monne M, Ouchi D, Piccolo Ferreira F, Malchair P, Videla S, Garcia Garcia V, Ruiz-Comellas A, Ramirez-Morros A, Rodriguez Codina J, Amado Simon R, Grifols JR, Blanco J, Blanco I, Ara J, Bassat Q, Clotet B, Baro B, Troxel A, Zwaginga JJ, Mitja O, Rijnders BJA; CoV-Early study group; COnV-ert study group. Prospective individual patient data meta-analysis of two randomized trials on convalescent plasma for COVID-19 outpatients. Nat Commun. 2022 May 11;13(1):2583. doi: 10.1038/s41467-022-29911-3. PMID 35546145
- [Derived] Alemany A, Millat-Martinez P, Corbacho-Monne M, Malchair P, Ouchi D, Ruiz-Comellas A, Ramirez-Morros A, Rodriguez Codina J, Amado Simon R, Videla S, Costes G, Capdevila-Jauregui M, Torrano-Soler P, San Jose A, Bonet Papell G, Puig J, Otero A, Ruibal Suarez JC, Zarauza Pellejero A, Llopis Roca F, Rodriguez Cortez O, Garcia Garcia V, Vidal-Alaball J, Millan A, Contreras E, Grifols JR, Ancochea A, Galvan-Femenia I, Piccolo Ferreira F, Bonet M, Cantoni J, Prat N, Ara J, Forcada Arcarons A, Farre M, Pradenas E, Blanco J, Angel Rodriguez-Arias M, Fernandez Rivas G, Marks M, Bassat Q, Blanco I, Baro B, Clotet B, Mitja O; CONV-ERT Group. High-titre methylene blue-treated convalescent plasma as an early treatment for outpatients with COVID-19: a randomised, placebo-controlled trial. Lancet Respir Med. 2022 Mar;10(3):278-288. doi: 10.1016/S2213-2600(21)00545-2. Epub 2022 Feb 9. PMID 35150610